CLINICAL TRIAL: NCT00727935
Title: Comparison Of The Analgesia Obtained By Infiltration Of Lidocaïne 1% And Ropivacaïne 0,75% Versus Placebo For The Joinings Of Episiotomies Among Parturients Under Epidural Analgesia
Brief Title: Comparison Of The Analgesia Obtained By Infiltration For The Joinings Of Episiotomies (Liropep)
Acronym: LiRoPep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU P 2006-03
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Parturients; Childbirth
Keywords: Women; parturients; with; realization; episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lidocaïne
Drug: Ropivacaïne
Drug: Placebo

SUMMARY:
Lateral episiotomy is a current care practiced with childbirth room. One of the problems encountered with this surgical act is the residual pain on perineal scar level. Maximal during the first 24 hours, this pain can persist several days or several weeks hampering to variable degrees a normal recovery of autonomy and comfort of life. Some studies have shown the interest of ropivacaine, local anaesthetic with a long action's duration for proctologic surgeries and for the cure of inguinal hernia. A recent study shown the ropivacaine perineal infiltration used prior perineorrhaphy allows an absence of post-partum pain for 24 to 27% of cases and a first analgesics request delayed to ten hours.

Methodology: 165 parturients having an epidural analgesia and an episiotomy were enrolled. The perineal infiltration was randomized according to 3 equal groups (placebo, ropivacaine 0,75%, lidocaine 1%) and realised prior perineorrhaphy. then The parturient were followed during the 24 first hours. This study was designed as double blind and the study conduct was standardized in order to get only variable such as the episiotomy infiltration.

ELIGIBILITY:
Pre-inclusion criteria :

* Assent of participation in the study signed
* Major parturient (> 18 years) in the course of work in room of childbirth
* Mono-foetal pregnancy
* Presentation at the top

Inclusion Criteria:

* Checking of the criteria of pre-inclusion
* Oral confirmation of the assent of the patient
* ASA 1 or 2
* Childbirth by low way
* Patient having an epidural analgesia
* Patient having an episiotomy
* Counter-indication with the ropivacaïne

Pre-exclusion criteria :

* Absence of signed assent of participation in the study
* Counter indication with the lidocaïne
* General counter-indications suitable for the epidural anaesthesia , independently of the local anaesthetic used
* Counter-indications with the infiltration: patient under anticoagulants, coagulopathy
* Allergy to the lidocaine or the ropivacaine
* Allergy to the one of analgesics per bones used in the assumption of responsibility of routine
* Severe insufficiency hepatic and/or renal and/or ulcerates gastro-duodénal (in the case of anti-inflammatory drug regulation not steroid during the postpartum)
* Minor
* Major protected within the meaning of the law Huriet
* Patient during one time of exclusion following another biomedical study

Exclusion Criteria:

* Absence of oral confirmation of the assent of the patient
* Infection or ignition of the point of puncture
* Analgesia epidural not functional
* Dural breach
* Appearance of ascribable side effects to only the anaesthetic buildings at the time of epidural analgesia
* Median Episiotomy (increased risk of lesions of the sphincter)
* Need for an instrumentation at the time of expulsion
* Haemorrhage of the delivery requiring a blood transfusion and/or general anaesthesia in urgency with surgical operation for haemostasis

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time between the infiltration of the local anaesthetic and the first analgesics catch per os, which is managed when the level of pain evaluated by EVA is higher than 30 mm | 1 year

SECONDARY OUTCOMES:
To compare between the 3 groups the mean level of the pain during the first 24 hours following the joining of the episiotomy, measured by EVA | 24 hours
To compare between the 3 groups the analgesics overall consumption per os during the first 24 hours following the joining of the episiotomy | 24 hours
To compare between the 3 groups the total cost of the analgesics consumption (local anaesthetic employed and analgesics per bone) during the first 24 hours following the joining of the episiotomy | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Colbus, MD, Principal Investigator — Centre Hospitalier Universitaire Angers
Locations (1):
- Centre Hospitalier Universitaire, Angers, Pays de la Loire Region, France